CLINICAL TRIAL: NCT03329690
Title: A Phase 2, Multicenter, Open-label Study of DS-8201a in Subjects With HER2-expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: DS-8201a in Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Gastric Cancer [DESTINY-Gastric01]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-J202; 173727 (Registry Identifier: JAPIC CTI); DESTINY-G01 (Other: Daiichi Sankyo and AstraZeneca)
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2020-11-27 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Neoplasm, Gastrointestinal
Keywords: Adenocarcinoma Metastatic; Adenocarcinoma of the Stomach; Adenocarcinoma of the Gastroesophageal Junction; HER2 Overexpression; Adenocarcinoma, Locally Advanced; DESTINY - Gastric 01
MeSH Terms: conditions — Gastrointestinal Neoplasms; Adenocarcinoma | interventions — trastuzumab deruxtecan; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two randomized investigative arms will run in parallel (DS-8201a and Physician's Choice), with participants who have disease progression after two previous regimens.
  Two non-randomized exploratory arms will run with HER2 treatment-naive participants.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Parallel: DS-8201a (Experimental): Participants with HER2-overexpressing (IHC 3+ or IHC 2+/ISH+) advanced gastric or gastroesophageal junction adenocarcinoma, whose disease has progressed on two prior regimens, will receive DS-8201a once every 3 weeks.
  Interventions: Drug: DS-8201a
- Parallel: Physician's Choice (Active Comparator): Participants with HER2-overexpressing (IHC 3+ or IHC 2+/ISH+) advanced gastric or gastroesophageal junction adenocarcinoma, whose disease has progressed on two prior regimens, will receive monotherapy prescribed by the physician before enrollment.
  Interventions: Drug: Physician's Choice
- Exploratory: Naïve HER2 IHC 2+/ISH- (Other): A maximum of 20 non-randomized participants with HER2 IHC 2+/ISH- advanced gastric or gastroesophageal junction adenocarcinoma will receive DS-8201a once every three weeks.
  Interventions: Drug: DS-8201a
- Exploratory: Naïve HER2 IHC 1+ (Other): A maximum of 20 non-randomized patients with HER2 IHC 1+ advanced gastric or gastroesophageal junction adenocarcinoma will receive DS-8201a once every 3 weeks.
  Interventions: Drug: DS-8201a

INTERVENTIONS:
Drug: DS-8201a — DS-8201a is comprised of an antibody component conjoined to a drug component in a lyophilized powder, which is made into solution for intravenous administration.
  Other Names: Experimental product
  Arms: Exploratory: Naïve HER2 IHC 1+; Exploratory: Naïve HER2 IHC 2+/ISH-; Parallel: DS-8201a
Drug: Physician's Choice — Either:
  Irinotecan monotherapy (Starting dosage and usage is 150 mg/m2 biweekly, with dose reduction permitted)
  Paclitaxel monotherapy (Starting dosage and usage is 80 mg/m2 weekly, with dose reduction permitted)
  Other Names: Standard of Care
  Arms: Parallel: Physician's Choice

SUMMARY:
The primary purpose of this trial is to compare the efficacy and safety of DS-8201a and physician's choice treatment in HER2-overexpressing advanced gastric or gastroesophageal junction adenocarcinoma patients who have progressed on two prior treatment regimens including fluoropyrimidine agent, platinum agent, and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Has a pathologically documented locally advanced or metastatic adenocarcinoma of gastric or gastroesophageal junction
2. Progression on and after at least 2 prior regimens
3. Has an adequate tumor sample
4. Has measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1

Exclusion Criteria:

1. Has a medical history of myocardial infarction, symptomatic congestive heart failure (CHF) (NYHA classes II-IV), unstable angina or serious cardiac arrhythmia
2. Has a QTc prolongation to > 450 millisecond (ms) in males and > 470 ms in females
3. Has a medical history of clinically significant lung disease
4. Is suspected to have certain other protocol-defined diseases based on imaging at screening period
5. Has history of any disease, metastatic condition, drug/medication use or other condition that might, per protocol or in the opinion of the investigator, compromise:

   1. safety or well-being of the participant or offspring
   2. safety of study staff
   3. analysis of results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (66):
- Japan (48):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Japan Community Health Care Organization Kyushu Hospital, Kitakyushu, Fukuoka
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Kure Medical Center, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagawa University Hospital, Kita, Kagawa-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - The Kitasato Institute Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Japanese Red Cross Kyoto Daini Hospital, Kamigyō-ku, Kyoto
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Osaki Citizen Hospital, Ōsaki, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - Toyonaka Municipal Hospital, Toyonaka, Osaka
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Tokyo Metropolitan Komagome Hospital, Bunkyō-Ku, Tokyo
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-Ku, Tokyo
  - Showa University Koto Toyosu Hospital, Koto-Ku, Tokyo
  - Toranomon Hospital, Minato-Ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Fukui Prefectural Hospital, Fukui
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima City Asa Citizens Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Kochi Health Sciences Center, Kochi
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Local Incorporated Administrative Agency Osaka City Hospital Organization Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Osaka General Medical Center, Osaka
  - Kindai University Hospital, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka
  - Keio University Hospital, Tokyo
- South Korea (18):
  - National Cancer Center, Ilsan, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center, Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Result] Shitara K, Bang YJ, Iwasa S, Sugimoto N, Ryu MH, Sakai D, Chung HC, Kawakami H, Yabusaki H, Lee J, Saito K, Kawaguchi Y, Kamio T, Kojima A, Sugihara M, Yamaguchi K; DESTINY-Gastric01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Gastric Cancer. N Engl J Med. 2020 Jun 18;382(25):2419-2430. doi: 10.1056/NEJMoa2004413. Epub 2020 May 29. PMID 32469182
- [Derived] Yamaguchi K, Bang YJ, Iwasa S, Sugimoto N, Ryu MH, Sakai D, Chung HC, Kawakami H, Yabusaki H, Lee J, Shimoyama T, Lee KW, Saito K, Kawaguchi Y, Kamio T, Kojima A, Sugihara M, Shitara K. Trastuzumab Deruxtecan in Anti-Human Epidermal Growth Factor Receptor 2 Treatment-Naive Patients With Human Epidermal Growth Factor Receptor 2-Low Gastric or Gastroesophageal Junction Adenocarcinoma: Exploratory Cohort Results in a Phase II Trial. J Clin Oncol. 2023 Feb 1;41(4):816-825. doi: 10.1200/JCO.22.00575. Epub 2022 Nov 15. PMID 36379002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the Primary Cohort, a total of 188 participants who met all inclusion criteria and no exclusion criteria were enrolled and randomized to treatment. In the Exploratory Cohorts, a total of 45 non-randomized participants were enrolled and 44 patients received treatment. Study participants for all cohorts were enrolled at clinic sites in South Korea and Japan. Participants took part of the study from November 2, 2017 to Data Cut-Off (DCO) date of December 11, 2020.
Pre-assignment Details: In the Primary Cohort, participants with HER2 overexpressing gastric of GEJ adenocarcinoma were randomized (2:1) to either DS-8201a or physician's choice (irinotecan or paclitaxel). In the Exploratory Cohorts, participants with HER2 IHC 2+/ISH negative advanced gastric or GEJ adenocarcinoma who were naïve to HER2 treatment received DS-8201a.
Groups:
- DS-8201a: Participants with HER2-overexpressing (IHC 3+ or IHC 2+/ISH+) advanced gastric or gastroesophageal junction adenocarcinoma, whose disease had progressed on two prior regimens, were randomized to receive DS-8201a once every 3 weeks.
- Physician's Choice Irinotecan: Participants with HER2-overexpressing (IHC 3+ or IHC 2+/ISH+) advanced gastric or gastroesophageal junction adenocarcinoma, whose disease had progressed on two prior regimens, were randomized to receive irinotecan monotherapy as prescribed by the physician before enrollment.
- Physician's Choice Paclitaxel: Participants with HER2-overexpressing (IHC 3+ or IHC 2+/ISH+) advanced gastric or gastroesophageal junction adenocarcinoma, whose disease had progressed on two prior regimens, were randomized to receive paclitaxel monotherapy as prescribed by the physician before enrollment.
- Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a: Non-randomized participants with HER2 IHC 2+/ISH- advanced gastric or gastroesophageal junction adenocarcinoma who received DS-8201a once every three weeks.
- Exploratory: Naïve HER2 IHC 1+, DS-8201a: Non-randomized participants with HER2 IHC 1+ advanced gastric or gastroesophageal junction adenocarcinoma who received DS-8201a once every 3 weeks.
Period: Overall Study
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Started | 126 | 55 | 7 | 21 | 24
Received Treatment | 125 | 55 | 7 | 20 | 24
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 126 | 55 | 7 | 21 | 24
Not completed — Progressive disease per RECIST | 85 | 44 | 6 | 16 | 20
Not completed — Clinical progression | 7 | 4 | 1 | 1 | 1
Not completed — Adverse Event | 22 | 4 | 0 | 1 | 2
Not completed — Death | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 1
Not completed — Miscellaneous | 6 | 0 | 0 | 0 | 0
Not completed — Did not receive treatment | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline and demographic characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a | Total
Number analyzed (Participants) | 125 | 55 | 7 | 20 | 24 | 231
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 24 | 3 | 11 | 17 | 110
  >=65 years | 70 | 31 | 4 | 9 | 7 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.36) | 64.9 (10.54) | 63.4 (8.96) | 62.5 (10.87) | 55.5 (12.12) | 63.3 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 13 | 2 | 4 | 7 | 56
  Male | 95 | 42 | 5 | 16 | 17 | 175
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 125 | 55 | 7 | 20 | 24 | 231
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 26 | 11 | 1 | 4 | 5 | 47
  Japan | 99 | 44 | 6 | 16 | 19 | 184

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Rate Based on Independent Central Review Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Intent-to-Treat Analysis Set)
Description: The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR), assessed by independent central imaging review (ICR) based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Unconfirmed ORR (not confirmed by ICR) and confirmed ORR (confirmed by ICR) are reported.
Time Frame: Baseline to date of first documented objective response (CR or PR), up to 36 months postdose
Population: Objective response rate was assessed in the Primary Cohort in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Physician's Choice Overall: Participants with HER2-overexpressing (IHC 3+ or IHC 2+/ISH+) advanced gastric or gastroesophageal junction adenocarcinoma, whose disease had progressed on two prior regimens, were randomized to receive either irinotecan or paclitaxel monotherapy as prescribed by the physician before enrollment.
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall
Number analyzed (Participants) | 126 | 55 | 7 | 62
Participants
  Unconfirmed ORR, 25 months (DCO: Nov 8, 2019) | 61 | 7 | 1 | 8
  Unconfirmed ORR, 36 months (DCO: Dec 11, 2020) | 61 | 7 | 1 | 8
  Confirmed ORR, 25 months (DCO: Nov 8, 2019) | 51 | 6 | 1 | 7
  Confirmed ORR, 36 months (DCO: Dec 11, 2020) | 50 | 6 | 1 | 7
Statistical Analysis 1: Comparison: DS-8201a vs Physician's Choice Overall; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; CMH test with region as a stratification factor

2. Primary Outcome: Percentage of Participants With Best Overall Response Based on Independent Central Review Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Intent-to-Treat Analysis Set)
Description: The best overall response is the best overall response (BOR) recorded from the start of the study treatment until the end of treatment and includes complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) and not evaluable (NE) as assessed by independent central imaging review (ICR) based on RECIST version 1.1. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. Unconfirmed BOR (not confirmed by ICR) and confirmed BOR (confirmed by ICR) are reported.
Time Frame: Baseline to date of first documented objective response, up to 36 months postdose
Population: Best overall response was assessed in the Primary Cohort in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall
Number analyzed (Participants) | 126 | 55 | 7 | 62
Participants
  Unconfirmed Complete response (CR), 25 months (DCO: Nov 8, 2019) | 11 | 0 | 0 | 0
  Unconfirmed Complete response (CR), 36 months (DCO: Dec 11, 2020) | 10 | 0 | 0 | 0
  Unconfirmed Partial response (PR), 25 months (DCO: Nov 8, 2019) | 50 | 7 | 1 | 8
  Unconfirmed Partial response (PR), 36 months (DCO: Dec 11, 2020) | 51 | 7 | 1 | 8
  Unconfirmed Stable disease (SD), 25 months (DCO: Nov 8, 2019) | 46 | 27 | 3 | 30
  Unconfirmed Stable disease (SD), 36 months (DCO: Dec 11, 2020) | 47 | 27 | 3 | 30
  Unconfirmed Progressive disease (PD), 25 months (DCO: Nov 8, 2019) | 15 | 18 | 0 | 18
  Unconfirmed Progressive disease (PD), 36 months (DCO: Dec 11, 2020) | 15 | 18 | 0 | 18
  Unconfirmed Not evaluable (NE), 25 months (DCO: Nov 8, 2019) | 4 | 3 | 3 | 6
  Unconfirmed Not evaluable (NE), 36 months (DCO: Dec 11, 2020) | 3 | 3 | 3 | 6
  Confirmed Complete response (CR), 25 months (DCO: Nov 8, 2019) | 10 | 0 | 0 | 0
  Confirmed Complete response (CR), 36 months (DCO: Dec 11, 2020) | 9 | 0 | 0 | 0
  Confirmed Partial response (PR), 25 months (DCO: Nov 8, 2019) | 41 | 6 | 1 | 7
  Confirmed Partial response (PR), 36 months (DCO: Dec 11, 2020) | 41 | 6 | 1 | 7
  Confirmed Stable disease (SD), 25 months (DCO: Nov 8, 2019) | 55 | 28 | 3 | 31
  Confirmed Stable disease (SD), 36 months (DCO: Dec 11, 2020) | 57 | 28 | 3 | 31
  Confirmed Progressive disease (PD), 25 months (DCO: Nov 8, 2019) | 15 | 18 | 0 | 18
  Confirmed Progressive disease (PD), 36 months (DCO: Dec 11, 2020) | 15 | 18 | 0 | 18
  Confirmed Not evaluable (NE), 25 months (DCO: Nov 8, 2019) | 5 | 3 | 3 | 6
  Confirmed Not evaluable (NE), 36 months (DCO: Dec 11, 2020) | 4 | 3 | 3 | 6

3. Secondary Outcome: Overall Survival Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Intent-to-Treat Analysis Set)
Description: Duration of survival follow-up (months) was defined as the date of last contact - date of randomization/ registration + 1.Overall Survival (OS) was defined as the time from the date of randomization (the date of the registration for the Exploratory Cohorts) to the date of death due to any cause.
Time Frame: From the date of randomization to the date of death (due to any cause), up to 36 months postdose
Population: Duration of survival and overall survival were assessed in the Intent-to-Treat Analysis Set.
Measure: Median (Full Range); unit: months
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 126 | 55 | 7 | 62 | 21 | 22
months
  Duration of survival follow up, 25 months (DCO: Nov 8, 2019) | 8.0 [0.4 to 23.1] | 7.1 [0.3 to 20.3] | 5.5 [2.0 to 14.3] | 7.0 [0.3 to 20.3] | 7.3 [0.2 to 19.6] | 8.4 [1.8 to 14.8]
  Duration of survival follow up, 36 months (DCO: Dec 11, 2020) | 12.3 [0.4 to 33.2] | 8.4 [0.3 to 29.3] | 14.3 [2.0 to 22.1] | 8.5 [0.3 to 29.3] | 7.3 [0.2 to 27.7] | 8.5 [1.8 to 23.1]
  Overall survival, 25 months (DCO: Nov 8, 2019) | 12.5 [0.4 to 23.1] | 8.4 [0.3 to 20.3] | 14.3 [2.0 to 14.3] | 8.4 [0.3 to 20.3] | 7.8 [0.2 to 19.6] | 8.5 [1.8 to 14.8]
  Overall survival, 36 months (DCO: Dec 11, 2020) | 12.6 [0.4 to 33.2] | 8.6 [0.3 to 29.3] | 14.3 [2.0 to 22.1] | 8.9 [0.3 to 29.3] | 7.8 [0.2 to 27.7] | 8.5 [1.8 to 23.1]

4. Secondary Outcome: Progression-Free Survival Based on Independent Central Review Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Intent-to-Treat Analysis Set)
Description: Progression-free survival (PFS) was defined as the time from the date of randomization (the date of the registration for the Exploratory Cohorts) to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From the date of randomization to the first documented disease progression or date of death (whichever occurs first), up to 36 months postdose
Population: Progression-free survival (PFS) was assessed in the Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 126 | 55 | 7 | 62 | 21 | 22
months
  PFS, 25 months (DCO: Nov 8, 2019) | 5.6 [4.3 to 6.9] | 2.8 [2.0 to 4.3] | 4.9 [2.0 to NA] — Missing upper limit was not calculable due to right censored data; last timepoint censored and estimate is infinity. | 3.5 [2.0 to 4.3] | 4.4 [2.7 to 7.1] | 2.8 [1.5 to 4.3]
  PFS, 36 months (DCO: Dec 11, 2020) | 5.6 [4.3 to 6.9] | 2.8 [2.0 to 4.3] | 4.9 [2.0 to NA] — Missing upper limit was not calculable due to right censored data; last timepoint censored and estimate is infinity. | 3.5 [2.0 to 4.3] | 4.4 [2.7 to 7.1] | 2.8 [1.5 to 4.3]

5. Secondary Outcome: Duration of Response Based on Independent Central Review Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Full Analysis Set)
Description: Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR was measured for responding subjects (PR or CR) only.
Time Frame: From the date of first objective response (CR or PR) to the date of first documentation of PD or death (whichever occurs first), up to 36 months postdose
Population: Duration of response (DOR) was assessed in the Full Analysis Set.
Measure: Median (Full Range); unit: months
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 61 | 7 | 1 | 8 | 7 | 4
months
  Unconfirmed Duration of response (DOR), 25 months (DCO: Nov 8, 2019) | 8.4 [0 to 21.0] | 4.1 [0 to 4.9] | 3.9 [3.9 to 3.9] | 3.9 [0 to 4.9] | 6.8 [1.4 to 9.7] | 7.1 [1.4 to 12.5]
  Unconfirmed Duration of response (DOR), 36 months (DCO: Dec 11, 2020) | 11.3 [0 to 29.1] | 4.1 [0 to 4.9] | 3.9 [3.9 to 3.9] | 3.9 [0 to 4.9] | 6.8 [1.4 to 12.5] | 5.8 [1.4 to 12.5]
  Confirmed Duration of response (DOR), 25 months (DCO: Nov 8, 2019): number analyzed (Participants) | 51 | 6 | 1 | 7 | 5 | 2
  Confirmed Duration of response (DOR), 25 months (DCO: Nov 8, 2019) | 11.3 [1.4 to 21.0] | 4.1 [1.4 to 4.9] | 3.9 [3.9 to 3.9] | 3.9 [1.4 to 4.9] | 7.6 [2.4 to 9.7] | 12.5 [8.1 to 12.5]
  Confirmed Duration of response (DOR), 36 months (DCO: Dec 11, 2020): number analyzed (Participants) | 50 | 6 | 1 | 7 | 5 | 2
  Confirmed Duration of response (DOR), 36 months (DCO: Dec 11, 2020) | 12.7 [1.4 to 29.1] | 4.1 [1.4 to 4.9] | 3.9 [3.9 to 3.9] | 3.9 [1.4 to 4.9] | 7.6 [2.4 to 12.5] | 11.2 [10.0 to 12.5]

6. Secondary Outcome: Disease Control Rate With and Without Confirmation by Independent Central Review Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Intent-to-Treat Analysis Set)
Description: Disease control rate (DCR) was defined as the sum of complete response (CR) rate, partial response (PR) rate, and stable disease (SD) rate. As per RECIST v1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Baseline to date of first documented objective response (CR, PR, and SD), up to 36 months postdose
Population: Disease control rate (DCR) was assessed in the Intent-to-Treat Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 126 | 55 | 7 | 62 | 21 | 22
Participants
  DCR, 25 months (DCO: Nov 8, 2019) | 107 | 34 | 4 | 38 | 17 | 15
  DCR, 36 months (DCO: Dec 11, 2020) | 108 | 34 | 4 | 38 | 17 | 15

7. Secondary Outcome: Objective Response Rate and Best Overall Response Based on Independent Central Review Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Intent-to-Treat Analysis Set)
Description: The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR), assessed by Independent Central Review (ICR) based on RECIST version 1.1. The best overall response is the best overall response (BOR) recorded from the start of the study treatment until the end of treatment and includes CR, PR, stable disease (SD), progressive disease (PD) and not evaluable (NE) as assessed by Investigator based on RECIST version 1.1. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (at least a 20% increase in the sum of diameters of target lesions). Confirmed ORR and BOR (confirmed by ICR) are reported.
Time Frame: From randomization to first documented objective response, up to 36 months postdose
Population: Best overall response was assessed in the Exploratory Cohorts in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 21 | 22
Participants
  Confirmed Objective response rate (ORR), 25 months (DCO: Nov 8, 2019) | 5 | 2
  Confirmed Objective response rate (ORR), 36 months (DCO: Dec 11, 2020) | 5 | 2
  Confirmed Complete response (CR), 25 months (DCO: Nov 8, 2019) | 0 | 0
  Confirmed Complete response (CR), 36 months (DCO: Dec 11, 2020) | 0 | 0
  Confirmed Partial response (PR), 25 months (DCO: Nov 8, 2019) | 5 | 2
  Confirmed Partial response (PR), 36 months (DCO: Dec 11, 2020) | 5 | 2
  Confirmed Stable disease (SD), 25 months (DCO: Nov 8, 2019) | 12 | 13
  Confirmed Stable disease (SD), 36 months (DCO: Dec 11, 2020) | 12 | 13
  Confirmed Progressive disease (PD), 25 months (DCO: Nov 8, 2019) | 3 | 6
  Confirmed Progressive disease (PD), 36 months (DCO: Dec 11, 2020) | 3 | 6
  Inevaluable, 25 months (DCO: Nov 8, 2019) | 1 | 1
  Inevaluable, 36 months (DCO: Dec 11, 2020) | 1 | 1

8. Secondary Outcome: Time to Treatment Failure Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Full Analysis Set)
Description: Time to treatment failure (TTF) was defined as the time from the date of randomization (the date of the registration for Exploratory Cohorts) to the earliest date of the first objective documentation of progressive disease (PD), death due to any cause, or treatment discontinuation.
Time Frame: From date of randomization to first documentation of PD, death due to any cause, or treatment discontinuation (whichever comes first), up to 36 months postdose
Population: Time to treatment failure (TTF) was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 55 | 7 | 62 | 20 | 22
months
  TTF, 25 months (DCO: Nov 8, 2019) | 4.2 [3.9 to 5.1] | 2.6 [1.6 to 2.8] | 2.9 [1.1 to 6.8] | 2.6 [1.6 to 2.8] | 3.7 [1.7 to 5.5] | 2.2 [1.4 to 3.0]
  TTF, 36 months (DCO: Dec 11, 2020) | 4.3 [3.9 to 5.4] | 2.6 [1.6 to 2.8] | 2.9 [1.1 to 6.8] | 2.6 [1.6 to 2.8] | 3.7 [1.7 to 5.5] | 2.2 [1.4 to 3.0]

9. Secondary Outcome: Objective Response Rate and Best Overall Response Based on Investigator Assessment Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Response Evaluable Set)
Description: The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR), assessed by Investigator based on RECIST version 1.1. The best overall response is the best overall response (BOR) recorded from the start of the study treatment until the end of treatment and includes CR, PR, stable disease (SD), progressive disease (PD) and not evaluable (NE) as assessed by Investigator based on RECIST version 1.1. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (at least a 20% increase in the sum of diameters of target lesions). Unconfirmed ORR and BOR (not confirmed by Investigator) and confirmed ORR and BOR (confirmed by Investigator) are reported.
Time Frame: From randomization to first documented objective response, up to 36 months postdose
Population: Objective response rate (ORR) and best overall response (BOR) were assessed in the Response Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 119 | 51 | 5 | 56 | 19 | 21
Participants
  Unconfirmed Objective response rate (ORR), 25 months (DCO: Nov 8, 2019) | 60 | 7 | 1 | 8 | 10 | 5
  Unconfirmed Objective response rate (ORR), 36 months (DCO: Dec 11, 2020) | 60 | 7 | 1 | 8 | 10 | 5
  Unconfirmed Complete response (CR), 25 months (DCO: Nov 8, 2019) | 4 | 0 | 0 | 0 | 0 | 0
  Unconfirmed Complete response (CR), 36 months (DCO: Dec 11, 2020) | 4 | 0 | 0 | 0 | 0 | 0
  Unconfirmed Partial response (PR), 25 months (DCO: Nov 8, 2019) | 56 | 7 | 1 | 8 | 10 | 5
  Unconfirmed Partial response (PR), 36 months (DCO: Dec 11, 2020) | 56 | 7 | 1 | 8 | 10 | 5
  Unconfirmed Stable disease (SD), 25 months (DCO: Nov 8, 2019) | 42 | 27 | 1 | 28 | 7 | 8
  Unconfirmed Stable disease (SD), 36 months (DCO: Dec 11, 2020) | 42 | 27 | 1 | 28 | 7 | 8
  Unconfirmed Progressive disease (PD), 25 months (DCO: Nov 8, 2019) | 15 | 15 | 2 | 17 | 2 | 8
  Unconfirmed Progressive disease (PD), 36 months (DCO: Dec 11, 2020) | 15 | 15 | 2 | 17 | 2 | 8
  Unconfirmed Not evaluable (NE), 25 months (DCO: Nov 8, 2019) | 2 | 2 | 1 | 3 | 0 | 0
  Unconfirmed Not evaluable (NE), 36 months (DCO: Dec 11, 2020) | 2 | 2 | 1 | 3 | 0 | 0
  Confirmed Objective response rate (ORR), 25 months (DCO: Nov 8, 2019) | 49 | 5 | 1 | 6 | 8 | 3
  Confirmed Objective response rate (ORR), 36 months (DCO: Dec 11, 2020) | 51 | 5 | 1 | 6 | 8 | 3
  Confirmed Complete response (CR), 25 months (DCO: Nov 8, 2019) | 3 | 0 | 0 | 0 | 0 | 0
  Confirmed Complete response (CR), 36 months (DCO: Dec 11, 2020) | 4 | 0 | 0 | 0 | 0 | 0
  Confirmed Partial response (PR), 25 months (DCO: Nov 8, 2019) | 46 | 5 | 1 | 6 | 8 | 3
  Confirmed Partial response (PR), 36 months (DCO: Dec 11, 2020) | 47 | 5 | 1 | 6 | 8 | 3
  Confirmed Stable disease (SD), 25 months (DCO: Nov 8, 2019) | 53 | 28 | 1 | 29 | 9 | 10
  Confirmed Stable disease (SD), 36 months (DCO: Dec 11, 2020) | 51 | 28 | 1 | 29 | 9 | 10
  Confirmed Progressive disease (PD), 25 months (DCO: Nov 8, 2019) | 15 | 16 | 2 | 18 | 2 | 8
  Confirmed Progressive disease (PD), 36 months (DCO: Dec 11, 2020) | 15 | 16 | 2 | 18 | 2 | 8
  Confirmed Not evaluable (NE), 25 months (DCO: Nov 8, 2019) | 2 | 2 | 1 | 3 | 0 | 0
  Confirmed Not evaluable (NE), 36 months (DCO: Dec 11, 2020) | 2 | 2 | 1 | 3 | 0 | 0

10. Secondary Outcome: Pharmacokinetic Parameter of Maximum Observed Serum Concentration (Cmax) and Trough Serum Concentration (Ctrough) of DS-8201a and Total Anti-HER2 Antibody Following Treatment With DS-8201a
Description: Blood samples for DS-8201a pharmacokinetic (PK) analysis were obtained at the specified timepoints. The maximum serum concentration (Cmax) and the trough serum concentration (Ctrough) of DS-8201a were assessed. These serum PK parameters for DS-8201a and total anti-HER2 antibody were estimated in each participant using standard noncompartmental methods.
Time Frame: Cycle 1 and 3, Day 1: predose, 4 hours (h), 7h postdose; Day 8, Day 15, and Day 22 postdose; Cycle 2, Day 1 and Day 22 postdose; Cycle 4, 6, and 8, Day 1 postdose (each cycle is 21 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DS-8201a | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 20 | 24
ug/mL
  Cmax: DS-8201a, Cycle 1 | 127 (28.4) | 119 (29.1) | 127 (24.5)
  Cmax: DS-8201a, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Cmax: DS-8201a, Cycle 3 | 137 (31.1) | 128 (25.6) | 123 (23.2)
  Cmax: Total Anti-HER2 antibody, Cycle 1 | 116 (30.6) | 105 (26.1) | 110 (19.6)
  Cmax: Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Cmax: Total Anti-HER2 antibody, Cycle 3 | 121 (28.4) | 115 (24.2) | 112 (21.9)
  Ctrough: DS-8201a, Cycle 1 | 5.56 (3.08) | 4.52 (2.42) | 9.51 (23.4)
  Ctrough: DS-8201a, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Ctrough: DS-8201a, Cycle 3 | 13.4 (17.3) | 8.84 (3.09) | 13.2 (18.6)
  Ctrough: Total Anti-HER2 antibody, Cycle 1 | 8.56 (8.60) | 5.33 (2.97) | 10.0 (20.5)
  Ctrough: Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Ctrough: Total Anti-HER2 antibody, Cycle 3 | 15.6 (13.6) | 12.2 (5.76) | 14.6 (17.6)

11. Secondary Outcome: Pharmacokinetic Parameter of Maximum Observed Serum Concentration (Cmax) and Trough Serum Concentration (Ctrough) of MAAA-1181 Following Treatment With DS-8201a
Description: Blood samples for DS-8201a pharmacokinetic (PK) analysis were obtained at the specified timepoints. The maximum serum concentration (Cmax) and the trough serum concentration (Ctrough) of DS-8201a were assessed. These serum PK parameters for MAAA-1181a were estimated in each participant using standard noncompartmental methods.
Time Frame: as for outcome 10
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-8201a | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 20 | 24
ng/mL
  Cmax: MAAA-1181a, Cycle 1 | 12.1 (4.79) | 13.3 (8.52) | 13.3 (7.37)
  Cmax: MAAA-1181a, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Cmax: MAAA-1181a, Cycle 3 | 9.08 (3.81) | 7.62 (1.86) | 9.83 (3.75)
  Ctrough: MAAA-1181a, Cycle 1 | 0.316 (0.294) | 0.290 (0.237) | 0.772 (2.28)
  Ctrough: MAAA-1181a Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Ctrough: MAAA-1181a Cycle 3 | 0.714 (2.19) | 0.378 (0.138) | 1.10 (1.95)

12. Secondary Outcome: Pharmacokinetic Parameters of Area Under the Concentration Versus-Time Curve of DS-8201a and Total Anti-HER2 Antibody Following Treatment With DS-8201a
Description: Blood samples for DS-8201a pharmacokinetic (PK) analysis were obtained at the specified timepoints. Area under the concentration versus time curve (AUC) from Time 0 to the Last Quantifiable Concentration (AUClast) and Area Under the Concentration versus-Time Curve up to 21 days (AUC21d) are reported. These serum PK parameters for DS-8201a and total anti-HER2 antibody were estimated in each participant using standard noncompartmental methods.
Time Frame: as for outcome 10
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set. No patient samples were collected or analyzed for AUClast DS-8201a and total anti-HER2 antibody for Cycle 3 as AUClast was planned to be assessed only for Cycle 1.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | DS-8201a | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 20 | 24
ug*d/mL
  AUClast: DS-8201a, Cycle 1 | 611 (150) | 572 (143) | 545 (160)
  AUClast: DS-8201a, Cycle 3: number analyzed (Participants) | 0 | 0 | 0
  AUClast: Total Anti-HER2 antibody, Cycle 1 | 667 (241) | 570 (126) | 547 (167)
  AUClast: Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 0 | 0 | 0
  AUC21d: DS-8201a, Cycle 1: number analyzed (Participants) | 124 | 20 | 23
  AUC21d: DS-8201a, Cycle 1 | 612 (150) | 572 (143) | 569 (114)
  AUC21d: DS-8201a, Cycle 3: number analyzed (Participants) | 66 | 10 | 10
  AUC21d: DS-8201a, Cycle 3 | 867 (213) | 746 (197) | 724 (71.9)
  AUC21d: Total Anti-HER2 antibody, Cycle 1: number analyzed (Participants) | 121 | 20 | 22
  AUC21d: Total Anti-HER2 antibody, Cycle 1 | 651 (210) | 570 (126) | 582 (104)
  AUC21d: Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 66 | 11 | 9
  AUC21d: Total Anti-HER2 antibody, Cycle 3 | 888 (244) | 775 (210) | 737 (110)

13. Secondary Outcome: Pharmacokinetic Parameters of Area Under the Concentration Versus-Time Curve of MAAA-1181 Following Treatment With DS-8201a
Description: Blood samples for DS-8201a pharmacokinetic (PK) analysis were obtained at the specified timepoints. Area under the concentration versus time curve (AUC) from Time 0 to the Last Quantifiable Concentration (AUClast) and Area Under the Concentration versus-Time Curve up to 21 days (AUC21d) are reported. These serum PK parameters for MAAA-1181a were estimated in each participant using standard noncompartmental methods.
Time Frame: as for outcome 10
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set. No patient samples were collected or analyzed for MAAA-1181a for Cycle 3 as AUClast was planned to be assessed only for Cycle 1.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | DS-8201a | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 20 | 24
ng*d/mL
  AUClast: MAAA-1181a, Cycle 1 | 46.7 (16.3) | 53.4 (42.7) | 44.5 (22.5)
  AUClast: MAAA-1181a, Cycle 3: number analyzed (Participants) | 0 | 0 | 0
  AUC21d: MAAA-1181a, Cycle 1: number analyzed (Participants) | 107 | 19 | 22
  AUC21d: MAAA-1181a, Cycle 1 | 46.4 (16.1) | 44.9 (20.1) | 44.5 (22.5)
  AUC21d: MAAA-1181a, Cycle 3: number analyzed (Participants) | 54 | 10 | 8
  AUC21d: MAAA-1181a, Cycle 3 | 42.0 (15.1) | 39.4 (8.36) | 44.6 (17.8)

14. Secondary Outcome: Pharmacokinetic Parameter of Time to Maximum Serum Concentration (Tmax) of DS-8201a, Total Anti-HER2 Antibody and MAAA-1181 Following Treatment With DS-8201a
Description: Blood samples for DS-8201a pharmacokinetic (PK) analysis were obtained at the specified timepoints. The time to maximum serum concentration (Tmax) of DS-8201a was assessed. This serum PK parameter for DS-8201a, total anti-HER2 antibody, and MAAA-1181a were estimated in each participant using standard noncompartmental methods.
Time Frame: as for outcome 10
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | DS-8201a | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 20 | 24
hours
  DS-8201a, Cycle 1 | 3.93 [0 to 7.15] | 3.90 [1.58 to 7.12] | 3.89 [1.53 to 7.08]
  DS-8201a, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  DS-8201a, Cycle 3 | 4.00 [0.58 to 7.25] | 4.00 [0.58 to 6.82] | 4.00 [0.68 to 7.02]
  Total Anti-HER2 antibody, Cycle 1 | 3.83 [0 to 7.15] | 3.83 [1.58 to 7.08] | 3.87 [1.53 to 7.08]
  Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  Total Anti-HER2 antibody, Cycle 3 | 3.98 [0.53 to 7.17] | 4.00 [0.57 to 6.83] | 3.75 [0.53 to 7.03]
  MAAA-1181a, Cycle 1 | 6.85 [3.75 to 7.25] | 6.83 [3.83 to 141.73] | 6.81 [3.83 to 7.08]
  MAAA-1181a, Cycle 3: number analyzed (Participants) | 69 | 11 | 11
  MAAA-1181a, Cycle 3 | 6.80 [3.78 to 7.25] | 6.82 [3.88 to 7.10] | 6.77 [3.98 to 7.07]

15. Secondary Outcome: Pharmacokinetic Parameter Terminal Elimination Half-life (t1/2) of DS-8201a, Total Anti-HER2 Antibody and MAAA-1181 Following Treatment With DS-8201a
Description: Blood samples for DS-8201a pharmacokinetic (PK) analysis were obtained at the specified timepoints. Terminal elimination half-life (t1/2) of DS-8201a was assessed. This serum PK parameter for DS-8201a, total anti-HER2 antibody, and MAAA-1181a were estimated in each participant using standard noncompartmental methods.
Time Frame: as for outcome 10
Population: Pharmacokinetic parameters were assessed in patients with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | DS-8201a | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 124 | 20 | 23
days
  DS-8201a, Cycle 1 | 5.77 (1.37) | 5.54 (1.08) | 5.52 (1.17)
  DS-8201a, Cycle 3: number analyzed (Participants) | 66 | 10 | 10
  DS-8201a, Cycle 3 | 7.46 (1.82) | 6.40 (1.00) | 6.35 (1.73)
  Total Anti-HER2 antibody, Cycle 1: number analyzed (Participants) | 121 | 20 | 22
  Total Anti-HER2 antibody, Cycle 1 | 6.20 (2.22) | 5.54 (1.01) | 5.65 (1.51)
  Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 66 | 11 | 9
  Total Anti-HER2 antibody, Cycle 3 | 8.00 (2.04) | 7.90 (2.10) | 6.17 (1.15)
  MAAA-1181a, Cycle 1: number analyzed (Participants) | 98 | 17 | 22
  MAAA-1181a, Cycle 1 | 5.50 (1.11) | 5.21 (0.939) | 5.61 (1.19)
  MAAA-1181a, Cycle 3: number analyzed (Participants) | 50 | 10 | 7
  MAAA-1181a, Cycle 3 | 7.01 (1.65) | 6.18 (1.02) | 5.80 (1.10)

16. Secondary Outcome: Overall Summary of Treatment-emergent Adverse Events (TEAEs) Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma. (Safety Analysis Set)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug. Serious adverse events (SAEs) with an onset or worsening 48 days or more after the last dose of study drug, if considered related to the study treatment, are also TEAEs.
Time Frame: Baseline up to 47 days after last dose, up to 36 months postdose
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 55 | 7 | 62 | 20 | 24
Participants
  Any TEAE, 25 months (DCO: Nov 8, 2019) | 125 | 54 | 7 | 61 | 20 | 24
  Any TEAE, 36 months (DCO: Dec 11, 2020) | 125 | 54 | 7 | 61 | 20 | 24
  Drug-related TEAEs, 25 months (DCO: Nov 8, 2019) | 122 | 51 | 5 | 56 | 19 | 24
  Drug-related TEAEs, 36 months (DCO: Dec 11, 2020) | 122 | 51 | 5 | 56 | 19 | 24
  Serious TEAEs, 25 months (DCO: Nov 8, 2019) | 55 | 14 | 1 | 15 | 6 | 11
  Serious TEAEs, 36 months (DCO: Dec 11, 2020) | 58 | 15 | 1 | 16 | 6 | 11
  Drug-related serious TEAEs, 25 months (DCO: Nov 8, 2019) | 27 | 5 | 0 | 5 | 1 | 6
  Drug-related serious TEAEs, 36 months (DCO: Dec 11, 2020) | 31 | 5 | 0 | 5 | 1 | 6
  TEAEs associated with drug withdrawn, 25 months (DCO: Nov 8, 2019) | 19 | 4 | 0 | 4 | 2 | 1
  TEAEs associated with drug withdrawn, 36 months (DCO: Dec 11, 2020) | 23 | 4 | 0 | 4 | 2 | 1
  Drug-related TEAEs associated with drug withdrawn, 25 months (DCO: Nov 8, 2019) | 12 | 3 | 0 | 3 | 1 | 0
  Drug-related TEAEs associated with drug withdrawn, 36 months (DCO: Dec 11, 2020) | 15 | 3 | 0 | 3 | 1 | 0
  TEAEs associated with dose reduced, 25 months (DCO: Nov 8, 2019) | 40 | 21 | 0 | 21 | 6 | 8
  TEAEs associated with dose reduced, 36 months (DCO: Dec 11, 2020) | 40 | 21 | 0 | 21 | 6 | 8
  Drug-related TEAEs associated with dose reduced, 25 months (DCO: Nov 8, 2019) | 38 | 21 | 0 | 21 | 6 | 7
  Drug-related TEAEs associated with dose reduced, 36 months (DCO: Dec 11, 2020) | 38 | 21 | 0 | 21 | 6 | 7
  TEAEs associated with drug interrupted, 25 months (DCO: Nov 8, 2019) | 78 | 20 | 3 | 23 | 8 | 10
  TEAEs associated with drug interrupted, 36 months (DCO: Dec 11, 2020) | 79 | 20 | 3 | 23 | 8 | 10
  Drug-related TEAE associated with drug interrupted, 25 months (DCO: Nov 8, 2019) | 64 | 17 | 2 | 19 | 7 | 10
  Drug-related TEAE associated with drug interrupted, 36 months (DCO: Dec 11, 2020) | 65 | 17 | 2 | 19 | 7 | 10
  TEAEs associated with death, 25 months (DCO: Nov 8, 2019) | 8 | 1 | 1 | 2 | 2 | 0
  TEAEs associated with death, 36 months (DCO: Dec 11, 2020) | 9 | 1 | 1 | 2 | 2 | 0

17. Secondary Outcome: Summary of Most Common Treatment-Emergent Adverse Events (TEAEs) ≥20% of Any Grade by Preferred Term Following Treatment With DS-8201a in Participants With HER2-Expressing Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (Safety Analysis Set)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug.
Time Frame: Baseline up to 47 days after last dose, up to 36 months postdose
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
Number analyzed (Participants) | 125 | 55 | 7 | 62 | 20 | 24
Participants
  Any TEAE, 25 months (DCO: Nov 8, 2019) | 125 | 54 | 7 | 61 | 20 | 24
  Any TEAE, 36 months (DCO: Dec 11, 2020) | 125 | 54 | 7 | 61 | 20 | 24
  Nausea, 25 months (DCO: Nov 8, 2019) | 79 | 27 | 2 | 29 | 11 | 19
  Nausea, 36 months (DCO: Dec 11, 2020) | 79 | 27 | 2 | 29 | 11 | 19
  Decreased appetite, 25 months (DCO: Nov 8, 2019) | 75 | 27 | 1 | 28 | 13 | 18
  Decreased appetite, 36 months (DCO: Dec 11, 2020) | 76 | 27 | 1 | 28 | 13 | 18
  Neutrophil count decreased, 25 months (DCO: Nov 8, 2019) | 77 | 18 | 3 | 21 | 8 | 12
  Neutrophil count decreased, 36 months (DCO: Dec 11, 2020) | 79 | 18 | 3 | 21 | 8 | 12
  Anaemia, 25 months (DCO: Nov 8, 2019) | 71 | 17 | 2 | 19 | 10 | 10
  Anaemia, 36 months (DCO: Dec 11, 2020) | 71 | 17 | 2 | 19 | 10 | 11
  White blood cell count decreased, 25 months (DCO: Nov 8, 2019) | 47 | 18 | 3 | 21 | 4 | 7
  White blood cell count decreased, 36 months (DCO: Dec 11, 2020) | 49 | 18 | 3 | 21 | 4 | 7
  Platelet count decreased, 25 months (DCO: Nov 8, 2019) | 47 | 4 | 0 | 4 | 3 | 7
  Platelet count decreased, 36 months (DCO: Dec 11, 2020) | 48 | 4 | 0 | 4 | 3 | 7
  Malaise, 25 months (DCO: Nov 8, 2019) | 43 | 9 | 1 | 10 | 4 | 9
  Malaise, 36 months (DCO: Dec 11, 2020) | 44 | 9 | 1 | 10 | 4 | 9
  Diarrhoea, 25 months (DCO: Nov 8, 2019) | 40 | 20 | 0 | 20 | 6 | 8
  Diarrhoea, 36 months (DCO: Dec 11, 2020) | 41 | 20 | 0 | 20 | 6 | 8
  Vomiting, 25 months (DCO: Nov 8, 2019) | 33 | 5 | 0 | 5 | 4 | 7
  Vomiting, 36 months (DCO: Dec 11, 2020) | 33 | 5 | 0 | 5 | 4 | 7
  Constipation, 25 months (DCO: Nov 8, 2019) | 30 | 13 | 1 | 14 | 5 | 5
  Constipation, 36 months (DCO: Dec 11, 2020) | 31 | 13 | 2 | 15 | 5 | 5
  Pyrexia, 25 months (DCO: Nov 8, 2019) | 30 | 8 | 2 | 10 | 3 | 6
  Pyrexia, 36 months (DCO: Dec 11, 2020) | 31 | 8 | 2 | 10 | 3 | 6
  Fatigue, 25 months (DCO: Nov 8, 2019) | 27 | 15 | 0 | 15 | 5 | 6
  Fatigue, 36 months (DCO: Dec 11, 2020) | 27 | 15 | 0 | 15 | 5 | 6
  Alopecia, 25 months (DCO: Nov 8, 2019) | 28 | 8 | 1 | 9 | 3 | 1
  Alopecia, 36 months (DCO: Dec 11, 2020) | 28 | 8 | 1 | 9 | 3 | 1
  Lymphocyte count decreased, 25 months (DCO: Nov 8, 2019) | 27 | 2 | 0 | 2 | 1 | 3
  Lymphocyte count decreased, 36 months (DCO: Dec 11, 2020) | 30 | 2 | 0 | 2 | 1 | 3
  Weight decreased, 25 months (DCO: Nov 8, 2019) | 17 | 5 | 0 | 5 | 4 | 7
  Weight decreased, 36 months (DCO: Dec 11, 2020) | 19 | 5 | 0 | 5 | 4 | 7
  Hypoalbuminaemia, 25 months (DCO: Nov 8, 2019) | 18 | 7 | 1 | 8 | 2 | 5
  Hypoalbuminaemia, 36 months (DCO: Dec 11, 2020) | 18 | 7 | 1 | 8 | 2 | 5
  Oedema peripheral, 25 months (DCO: Nov 8, 2019) | 13 | 0 | 0 | 0 | 4 | 1
  Oedema peripheral, 36 months (DCO: Dec 11, 2020) | 15 | 0 | 0 | 0 | 4 | 2
  Dysgeusia, 25 months (DCO: Nov 8, 2019) | 9 | 4 | 0 | 4 | 4 | 1
  Dysgeusia, 36 months (DCO: Dec 11, 2020) | 9 | 4 | 0 | 4 | 4 | 1
  Peripheral sensory neuropathy, 25 months (DCO: Nov 8, 2019) | 4 | 0 | 2 | 2 | 2 | 0
  Peripheral sensory neuropathy, 36 months (DCO: Dec 11, 2020) | 4 | 0 | 2 | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from baseline up to 47 days after last dose, up to 36 months postdose.
Description: A TEAE is defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug. Serious adverse events (SAEs) with an onset or worsening 48 days or more after the last dose of study drug, if considered related to the study treatment, are also TEAEs.
Arm/Group | DS-8201a | Physician's Choice Irinotecan | Physician's Choice Paclitaxel | Physician's Choice Overall | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a | Exploratory: Naïve HER2 IHC 1+, DS-8201a
All-Cause Mortality (participants affected / at risk) | 98/125 | 46/55 | 4/7 | 50/62 | 16/20 | 21/24
Serious Adverse Events (participants affected / at risk) | 58/125 | 15/55 | 1/7 | 16/62 | 6/20 | 11/24
Other Adverse Events (participants affected / at risk) | 125/125 | 54/55 | 7/7 | 61/62 | 20/20 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a (N=125) | Physician's Choice Irinotecan (N=55) | Physician's Choice Paclitaxel (N=7) | Physician's Choice Overall (N=62) | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a (N=20) | Exploratory: Naïve HER2 IHC 1+, DS-8201a (N=24)
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Device-related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Cholangitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1 | 0 | 0
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 0 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 1 | 0 | 1 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Gastric stenosis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 1 | 0 | 1 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 1 | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 3 | 2 | 0 | 2 | 2 | 0
Pyrexia (General disorders) | 3 | 1 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Condition aggravated (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a (N=125) | Physician's Choice Irinotecan (N=55) | Physician's Choice Paclitaxel (N=7) | Physician's Choice Overall (N=62) | Exploratory: Naïve HER2 IHC 2+/ISH-, DS-8201a (N=20) | Exploratory: Naïve HER2 IHC 1+, DS-8201a (N=24)
Nasopharyngitis (Infections and infestations) | 11 | 4 | 1 | 5 | 1 | 2
Pneumonia (Infections and infestations) | 7 | 1 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 1 | 2 | 0 | 1
Lung infection (Infections and infestations) | 6 | 0 | 0 | 0 | 2 | 1
Influenza (Infections and infestations) | 4 | 0 | 0 | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 0 | 3 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 3 | 2 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 71 | 17 | 2 | 19 | 10 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 0 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 76 | 27 | 1 | 28 | 13 | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 | 7 | 1 | 8 | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 4 | 0 | 4 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 8 | 2 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 3 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 4 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 3 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 11 | 4 | 1 | 5 | 2 | 1
Delirium (Psychiatric disorders) | 4 | 0 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 9 | 4 | 0 | 4 | 4 | 1
Dizziness (Nervous system disorders) | 5 | 3 | 0 | 3 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 0 | 4 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0 | 2 | 2 | 2 | 0
Cholinergic syndrome (Nervous system disorders) | 0 | 3 | 0 | 3 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 1
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 3
Hypertension (Vascular disorders) | 0 | 2 | 0 | 2 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0 | 6 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 79 | 27 | 2 | 29 | 11 | 19
Diarrhoea (Gastrointestinal disorders) | 41 | 20 | 0 | 20 | 6 | 8
Constipation (Gastrointestinal disorders) | 31 | 13 | 2 | 15 | 5 | 5
Vomiting (Gastrointestinal disorders) | 33 | 5 | 0 | 5 | 4 | 7
Abdominal pain (Gastrointestinal disorders) | 14 | 8 | 0 | 8 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 14 | 2 | 1 | 3 | 2 | 2
Ascites (Gastrointestinal disorders) | 8 | 2 | 0 | 2 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 0 | 2 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 0 | 3 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 1 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 10 | 1 | 0 | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 5 | 1 | 0 | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 8 | 1 | 9 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 2 | 0 | 2 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 0 | 1 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 1 | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 0
Malaise (General disorders) | 44 | 9 | 1 | 10 | 4 | 9
Fatigue (General disorders) | 27 | 15 | 0 | 15 | 5 | 6
Pyrexia (General disorders) | 31 | 8 | 2 | 10 | 3 | 6
Oedema peripheral (General disorders) | 15 | 0 | 0 | 0 | 4 | 2
Disease progression (General disorders) | 3 | 2 | 0 | 2 | 2 | 0
Asthenia (General disorders) | 1 | 3 | 0 | 3 | 0 | 2
Influenza-like illness (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 79 | 18 | 3 | 21 | 8 | 12
White blood cell count decreased (Investigations) | 49 | 18 | 3 | 21 | 4 | 7
Platelet count decreased (Investigations) | 48 | 4 | 0 | 4 | 3 | 7
Lymphocyte count decreased (Investigations) | 30 | 2 | 0 | 2 | 1 | 3
Weight decreased (Investigations) | 19 | 5 | 0 | 5 | 4 | 7
Aspartate aminotransferase increased (Investigations) | 12 | 3 | 0 | 3 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 11 | 1 | 1 | 2 | 1 | 4
Alanine aminotransferase increased (Investigations) | 9 | 3 | 0 | 3 | 1 | 0
Blood bilirubin increased (Investigations) | 10 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 6 | 0 | 6 | 2 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 0 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03329690/Prot_SAP_000.pdf